CLINICAL TRIAL: NCT03106064
Title: Independence in Self Care - A Program Focused on Nursing Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Cecília Maria Rodrigues, Nurse, Centro Hospitalar do Porto
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2016.037(032-DEFI/032-CES)
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Activities of Daily Living; Hospitalization; Nursing Care; Functional Impairment
MeSH Terms: interventions — Self Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Placebo Comparator): Intervention: Usual care
  Interventions: Other: Usual Care
- Intervention Group (Experimental): Intervention:Promoting independence in self-care
  Interventions: Behavioral: Promoting independence in self-care

INTERVENTIONS:
Behavioral: Promoting independence in self-care — The intervention will consist of an twice daily walking training, plus privileging trips to the toilet by walking (with support devices or with support from people) and all daytime meals seated (not in bed). Attending of the particular and unexplored characteristics of the proposed intervention, namely the use of the toilet and meals, the proposed intervention extends throughout the 24 hours of the day, seven days a week.
  Arms: Intervention Group
Other: Usual Care — Usual hospital care
  Arms: Usual Care Group

SUMMARY:
This study is a randomized clinical trial conducted in a medical ward of an acute 580-bedded teaching hospital. One hundred fifty-eight older acute medical patients will be blindly randomly allocated to the control group or intervention group. The intervention will consist of a twice daily walking training, plus privileging trips to the toilet by walking and all daytime meals seated. Differences between groups will be measured at baseline (admission) and discharge. As primary outcomes, we defined the length of stay and the independence level. The independence level will be assessed at baseline (admission) and discharge by two distinct methods: through the Barthel Index and the Patient Classification Systems(PCS).

DETAILED DESCRIPTION:
The intervention group will perform the training program while the control group will receive usual hospital care. As the study will be conducted in the same ward and due to the possible effect of subjects in the control group seeing subjects in the intervention group performing physical activity in addition to normal hospital care and because the service team itself may intervene involuntarily in the control group through increased activity, randomization will take place in a time dependent manner. Patients admitted for the first 12 weeks will be assigned to the control group. After these twelve weeks there will be a 3-week break and in the next 12 weeks (week 16 to 27) the admitted patients will be assigned to the intervention group. During the 3-week break, all members of the clinic staff will receive training on the intervention program.

All testing (at admission and discharge) will be performed in the same setting (Centro Hospitalar do Porto, Porto, Portugal) and by the same investigators.

Participants will include elderly people aged 65 years or older recruited from patients admitted into one of the three medical wards of the Centro Hospitalar do Porto (Porto, Portugal). Due to the length of the study it is possible a patient will be readmitted after participating in either the control or experimental group. To avoid this confounding variable, a study participant who is readmitted to the hospital during the course of the study will not be included in the study population a second time.

All clinical information will be obtained through direct observation of patients and consultation of medical records.

Interventions Usual care group (control) Participants assigned to the control group will receive usual hospital care, which includes physical rehabilitation when needed.

Intervention group (training) The intervention will consist of an twice daily walking training, plus privileging trips to the toilet by walking (with support devices or with support from people) and all daytime meals seated (not in bed). Attending of the particular and unexplored characteristics of the proposed intervention, namely the use of the toilet and meals, the proposed intervention extends throughout the 24 hours of the day, seven days a week. Therefore, it is an intervention that requires the alignment of the whole care team in its execution. The duration and quality of the training, planned for weeks 13 to 15, will be crucial to ensure the involvement of the whole team and the success of this study. We will re-organize the daily work of this particular service in order to focus nursing care on promoting independence in self-care.

Walk training will consist of walking as far as possible with or without assistance for 20 minutes. All training sessions will be individually monitored with a record of training completed compiled.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years or older.
* Able to ambulate, with or without personal/ technical assistance.
* Able to communicate.

Exclusion Criteria:

* Expected length of stay <72 hours
* Patients permanently bedridden prior to admission
* Any factor precluding performance of the physical training program. These factors include, but are not limited to the following:

  * Terminal illness.
  * Unstable cardiovascular disease or other medical condition.
  * Severe dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Independence level in self-care | The level of independence in self-care will be assessed at baseline (admission) and discharge through the Barthel Index
  Barthel Index: The sum-score ranges from 0 (totally dependent) to 100 (totally independent)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar do Porto - Departamento Qualidade, Porto, Portugal

REFERENCES:
- [Derived] Rodrigues C, Mendonca D, Martins MM. Effects of a nursing care program on functional outcomes in older acute medical in-patients: protocol for a randomized controlled trial. Porto Biomed J. 2018 Aug 1;4(2):e24. doi: 10.1016/j.pbj.0000000000000024. eCollection 2019 Mar-Apr. PMID 31595258